CLINICAL TRIAL: NCT01276561
Title: Single Incision Versus Standard Laparoscopic Splenectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09 09 196
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Hereditary Spherocytosis; Idiopathic Thrombocytopenic Purpura
Keywords: laparoscopy; splenectomy; single site; trial
MeSH Terms: conditions — Spherocytosis, Hereditary; Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Incision Splenectomy (Active Comparator): Patients will undergo splenectomy through a single incision in the umbilicus regardless of the technique or equipment used
  Interventions: Procedure: Single Incision Splenectomy
- Laparoscopic Splenectomy (Active Comparator): Patient will undergo standard laparoscopic splenectomy, port placement is surgeon dependent
  Interventions: Procedure: Laparoscopic Splenectomy

INTERVENTIONS:
Procedure: Single Incision Splenectomy — Patients will undergo laparoscopic splenectomy through a single incision
  Other Names: SILS
  Arms: Single Incision Splenectomy
Procedure: Laparoscopic Splenectomy — Patients will undergo laparoscopic splenectomy with 4 ports, placement is surgeon dependent
  Other Names: Standard
  Arms: Laparoscopic Splenectomy

SUMMARY:
This is a prospective trial of single incision versus standard 4-port laparoscopic splenectomy.

The hypothesis is that there may be a difference in wound infection rates, operative time, doses of analgesics post-operatively, and patient/parent perception of scars. However, the technical difficulty is considerable and the primary outcome is operative time which will be expressed in minutes.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial involving patients who present to the hospital with an indication for splenectomy. We will offer enrollment to several institutions provided they reach institutional approval.

This will be a definitive trial design. Based on our operative times with SILS compared with our recent experience in standard laparoscopy, a sample size of 30 patients will give us a power of 0.8 with an α of 0.05. Thus operative time is the primary outcome variable by definition. This is recorded and reported in MINUTES.

After the procedure, both groups will be managed in the same manner per routine care. They will be discharged when tolerating a regular diet and their pain is well-controlled on oral pain medication.

Secondary outcome measures include days in the hospital (measured in days), doses of analgesics (measured in doses) and perception of cosmesis as recorded by a scar assessment form which will be filled out by the patient and/or parents at 6 weeks and 6 months. This is a validated quality of life survey with 39 questions and each has 4 categories from best to worst.

ELIGIBILITY:
Inclusion Criteria:

* Need for splenectomy

Exclusion Criteria:

* Splenomegaly

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Operative time | 1 day
  operative time

SECONDARY OUTCOMES:
operative complications | 1 day
wound complications | 1 month
cosmesis | 6 months
length of stay | 1 week
operative difficulty | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No